CLINICAL TRIAL: NCT04685746
Title: BALANCED GROWTH: The Involvement of the Vestibular System in a Child's Cognitive and Motor Development
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201940165
Record Dates: First submitted 2020-12-11; First posted 2020-12-28 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Vestibular Disorder; Neurodevelopmental Disorders
MeSH Terms: conditions — Vestibular Diseases; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Typically developing school-aged children: Study group to achieve objective 1 and 2; control group to achieve objective 3 and 4 - Behavioural protocol: balanced growth protocol, consisting of audiovestibular, cognitive and motor assessments
  Interventions: Behavioral: Balanced Growth Protocol
- Vestibular-impaired school-aged children: Study group to achieve objective 3 - Behavioural protocol: balanced growth protocol, consisting of audiovestibular, cognitive and motor assessments
  Interventions: Behavioral: Balanced Growth Protocol
- Neurodevelopmental group (ADHD, ASD and/or DCD): Study group to achieve objective 4 - Behavioural protocol: balanced growth protocol, consisting of audiovestibular, cognitive and motor assessments
  Interventions: Behavioral: Balanced Growth Protocol

INTERVENTIONS:
Behavioral: Balanced Growth Protocol — Assessment of the Balanced Growth Protocol, consisting of audiovestibular testing, motor and cognitive tasks

SUMMARY:
When a vestibular dysfunction occurs at birth or in early stages of life, one might expect that this may have an enormous impact on a child's development. It is known that a severe congenital or early acquired vestibular deficit in children results in delayed psychomotor milestones. Later in life, children with a vestibular dysfunction may have difficulties with several balance tasks and additional cognitive, motor and/or psychosocial performances. While a few authors have suggested that there is indeed an influence of a vestibular dysfunction upon these different developmental domains (cognitive, motor, educational and psychosocial development), which can be supported by findings in clinical practice as well, literature concerning this topic remains fairly limited. On the other hand, several studies have shown that children with known difficulties in motor and/or cognitive functions have more difficulties in vestibular performances in comparison with their unaffected peers. Although more frequently discussed, the literature on this population is rather scarce too.

Therefore, the current project aims to investigate the relationship with and the involvement of the vestibular system in the motor and cognitive development of school-aged children.

DETAILED DESCRIPTION:
General goals

1. Developing and standardizing a sensitive and specific test protocol for the detection of vestibular, cognitive and/or motor dysfunctions in school-aged children.
2. Investigate the relationship with and the involvement of the vestibular system in the motor and cognitive development of typically developing school-aged children.
3. Investigating whether a vestibular dysfunction (with/without an additional auditory disease) has an impact on motor and/or cognitive performances in school-aged children.
4. Investigating if in children with a known neurodevelopmental disorder an (additional) underlying vestibular dysfunction can be identified.

ELIGIBILITY:
For typically developing children

Exclusion Criteria:

* Having a (permanent) hearing loss
* Having a (permanent) vestibular loss
* Having a motor dysfunction
* IQ < 70

For vestibular-impaired children

Inclusion Criteria:

* Recently (< 6 months) tested at the Ghent University Hospital
* Diagnosed with a vestibular impairment (= alteration on at least one of the vestibular function tests: caloric, rotatory chair, vHIT, cVEMP and/or oVEMP test)

For neurodevelopmental group

Inclusion Criteria:

• Diagnosed by a (neuro)psychiatric team with Autism Spectrum Disorder, Attention deficit/Hyperactivitiy Disorder and/or Developmental Coordination Disorder

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Typically developing children were used for establishing normative data of the protocol and to achieve objective 2 (convenience sampling; primary schools). Vestibular-impaired patients, established by extensive vestibular assessment for objective 3 (recruited at the Ghent University Hospital). The neurodevelopmental group was needed to establish objective 4 (recruited at schools for special education and/or care facilities).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
video Head Impulse Test gain (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the vHIT assessment (vestibular) which will take 5 minutes.
  Gain of the vestibulo-ocular reflex (high frequency function of the three semicircular canals)
video Head Impulse Test asymmetry (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the vHIT assessment (vestibular) which will take 5 minutes.
  Asymmetry of the vestibulo-ocular reflex between the left en right horizontal/anterior/posterior semicircular canals
video Head Impulse Test presence of saccades (overt/covert)(n) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the vHIT assessment (vestibular) which will take 5 minutes.
  Absolute amount of corrective saccades during head impulse testing
video Head Impulse Test presence of saccades (overt/covert)(% of the performed HITs) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the vHIT assessment (vestibular) which will take 5 minutes.
  Relative occurance of corrective saccades (with reference to the total amount of performed HITs) during head impulse testing
Rotatory chair gain (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the Rotatory chair assessment (vestibular) which will take 10 minutes.
  Gain of the vestibulo-ocular reflex (mid frequency function of the horizontal semicircular canals)
Rotatory chair phase (°) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the Rotatory chair assessment (vestibular) which will take 10 minutes.
  Phase lead between the eye and head velocity during rotatory chair testing
Rotatory chair asymmetry (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the Rotatory chair assessment (vestibular) which will take 10 minutes.
  Asymmetry of the vestibulo-ocular reflex between the left en right horizontal semicircular canal
Slow component velocity (SCV; °/s) in the culmination phase of each irrigation | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the caloric assessment (vestibular) which will take 15 minutes.
  The vestibulo-ocular reflex response (low frequency function of the horizontal semicircular canals)
Sum of all irrigations (°/s) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the caloric assessment (vestibular) which will take 15 minutes.
  The sum of the responses of the vestibulo-ocular reflex during the four irrigations
Unilateral weakness (UW; %) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the caloric assessment (vestibular) which will take 15 minutes.
  The asymmetry between the right and left horizontal semicircular canals (caloric testing)
Directional preponderance (DP; %) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the caloric assessment (vestibular) which will take 15 minutes.
  The asymmetry between nystagmus to the right vs to the left (caloric testing)
cVEMP: the absolute latencies of P1 and N1 (ms) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the cVEMP assessment (vestibular) which will take 5 minutes.
  Time between stimulation and onset of the response
cVEMP: rectified interpeak amplitude (µV) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the cVEMP assessment (vestibular) which will take 5 minutes.
  The amplitude of the cVEMP response
cVEMP: asymmetry ratio (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the cVEMP assessment (vestibular) which will take 5 minutes.
  The asymmetry between the right and left cVEMP response
oVEMP: the absolute latencies of N1 and P1 (ms) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the oVEMP assessment (vestibular) which will take 5 minutes.
  Time between stimulation and onset of the oVEMP response
oVEMP: interpeak amplitude (µV) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the oVEMP assessment (vestibular) which will take 5 minutes.
  The amplitude of the oVEMP response
oVEMP: asymmetry ratio (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the oVEMP assessment (vestibular) which will take 5 minutes.
  The asymmetry between the right and left oVEMP response
Movement assessment battery for children, Dutch version, 2nd edition (M ABC II NL): total score | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is part of the M ABC II NL assessment (motor) which will take 20 minutes.
  Total motor competence score of the participant (33 - max. 104, with a higher score indicating a higher motor competence)
Movement assessment battery for children, Dutch version, 2nd edition (M ABC II NL): subscale scores | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the M ABC II NL assessment (motor) which will take 20 minutes.
  Subscale scores of the M ABC II NL test battery
Movement assessment battery for children, Dutch version, 2nd edition (M ABC II NL): item scores | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the M ABC II NL assessment (motor) which will take 20 minutes.
  Item scores of the M ABC II NL test battery
Korpercoordination test fur kinder (KTK): raw scores (n) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the KTK assessment (motor) which will take 5 minutes.
  Amount of steps during the first subtest of the KTK (backward beam walking) (min. 0 - max. 72, with higher scores indicating better postural control during a dynamic balance task)
M CTSIB: the surface (mm²) of the confidence ellipse | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the M CTSIB assessment (motor) which will take 5 minutes.
  Confidence ellipse measured in millimeter² on force platform
M CTSIB: length covered by the consecutive center of pressure (COP) positions (mm) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the M CTSIB assessment (motor) which will take 5 minutes.
  Length of the COP measured in millimeter on force platform
M CTSIB: the mean velocity (mm/s) of the oscillations of the COP | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the M CTSIB assessment (motor) which will take 5 minutes.
  Mean celocity of the oscillations of the COP measured on force platform
M CTSIB: and the velocity variance (mm²/s²) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the M CTSIB assessment (motor) which will take 5 minutes.
  The oscillatory variance of the velocity of the COP measured on fore platform
Spatial span task: longest span (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The maximum number of squares that the subject correctly touched during the task
Spatial span task: amount of correct squares (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The absolute number of squares that the subject correctly touched during the task
Spatial span task: amount of correct squares (%) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The relative number of squares that the subject correctly touched during the task
Spatial span task: amount of incorrect squares (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The absolute number of incorrect squares that the subject touched during the task
Spatial span task: amount of incorrect squares (%) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The relative number of incorrect squares that the subject touched during the task
Spatial span task: amount of correct trials (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The absolute number of correct trials completed by the subject
Spatial span task: amount of correct trials (%) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The relative number of correct trials completed by the subject
Spatial span task: response rate (ms) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the spatial span assessment which will take 5 minutes.
  The response rate during each trial
Digit span task: longest span (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  The maximum number of digits that the subject correctly recalled during the task
Digit span task: amount of correct digits (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  cfr. spatial span
Digit span task: amount of correct digits (%) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  cfr. spatial span
Digit span task: amount of incorrect digits (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  cfr. spatial span
Digit span task: amount of incorrect digits (%) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  cfr. spatial span
Digit span task: number of correct trials (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  cfr. spatial span
Digit span task: number of correct trials (%) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  cfr. spatial span
Digit span task: response rate (ms) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the digit span assessment which will take 5 minutes.
  cfr. spatial span
Emotion recognition score (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the emotion recognition assessment which will take 5 minutes.
  Amount of correct recognized emotions per condition (NEPSY II NL)
Continuous performance task: omissions (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the attention assessment which will take 10 minutes.
  Amount of fails to press the button after the target appears
Continuous performance task: commissions (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the attention assessment which will take 10 minutes.
  "false alarm", when a participant presses the button for a non-target
Continuous performance task: total amount of errors (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the attention assessment which will take 10 minutes.
  Outcome 36 + 37
Continuous performance task: sustained attention | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the attention assessment which will take 10 minutes.
  Measured by calculating the change in hit and false alarm rates throughout the task
Continuous performance task: β | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the attention assessment which will take 10 minutes.
  Measure of impulsivity
Continuous performance task: d' | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the attention assessment which will take 10 minutes.
  Measure of visual selective attention; the probability of a hit vs a false alarm, taking into account the possibility of chance responding
Inhibition task: self-corrected errors naming (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of self-corrected errors during the condition "Naming" (NEPSY II NL)
Inhibition task: self-corrected errors inhibition (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of self-corrected errors during the condition "Inhibition" (NEPSY II NL)
Inhibition task: self-corrected errors switching (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of self-corrected errors during the condition "Switching" (NEPSY II NL)
Inhibition task: uncorrected errors naming (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of uncorrected errors during the condition "Naming" (NEPSY II NL)
Inhibition task: uncorrected errors inhibition (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of uncorrected errors during the condition "Inhibition" (NEPSY II NL)
Inhibition task: uncorrected errors switching (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of uncorrected errors during the condition "Switching" (NEPSY II NL)
Inhitbition task: total amount of errors naming (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of errors during the condition "Naming" (NEPSY II NL)
Inhitbition task: total amount of errors inhibition (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of errors during the condition "Inhibition" (NEPSY II NL)
Inhitbition task: total amount of errors switching (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Total amount of errors during the condition "Switching" (NEPSY II NL)
Inhitbition task: time naming (s) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Time needed to complete the condition "Naming" (NEPSY II NL)
Inhitbition task: time inhibition (s) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Time needed to complete the condition "Inhibition" (NEPSY II NL)
Inhitbition task: time switching (s) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the inhibition assessment which will take 10 minutes.
  Time needed to complete the condition "Switching" (NEPSY II NL)
Questionnaire Behaviour Rating Inventory of Executive Function (BRIEF) scores | This parameter will be assessed once during one of both testmoments (questionnaire for the parents), and is an outcome parameter of the executive function assessment which will take 10 minutes.
  The overall score and the subscores (n) of this validated questionnaire consisting of 75 items (3-point Likert scale) (min. 72 - max. 216, with higher scores indicating a higher level of executive functions)
Visual-Motor Integration (VMI) (Beery 6th edition): correct forms (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the visuo-motor assessment which will take 20 minutes.
  Total number of correct identified forms
Visual-Motor Integration (VMI) (Beery 6th edition): correct shapes (n) | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the visuo-motor assessment which will take 20 minutes.
  Total number of correctly completed shapes

SECONDARY OUTCOMES:
Score of the short version (4 subtest form) (Aubry & Bourdin, 2018) of the Wechsler Intelligence Scale for Children-VNL; WISC-V-NL | This parameter will be assessed once during one of both testmoments (the cognitive appointment), and is an outcome parameter of the intelligence assessment which will take 20 minutes.
  Estimated intelligence score based on the subtests "matrix reasoning", "similarities", "vocabulary", and "block design"; with a higher score indicating a higher intelligence quotient
Static visual acuity | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the ophtalmologic assessment which will take 5 minutes.
  The smallest optotype that can be correctly identified while the head is fixed
Dynamic visual acuity | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the ophtalmologic assessment which will take 5 minutes.
  The smallest optotype that can be correctly identified while moving the head
The difference between static visual acuity and dynamic visual acuity | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the ophtalmologic assessment which will take 5 minutes.
  This parameter results in the contribution of the vestibulo-ocular reflex during head movements
Tympanometry: middle ear pressure (daPa) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (tympanometry) which will take 1 minutes.
  Middle ear pressure of both ears
Tympanometry: static acoustic admitance (mmho) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (tympanometry) which will take 1 minutes.
  Static acoustic admitance (middle ear) of both ears
Tympanometry: ear canal volume (cm³) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (tympanometry) which will take 1 minutes.
  Ear canal volume of both ears
OAE measurement: stimulus stability (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (otoacoustic emissions) which will take 2 minutes.
  Stimulus stability during OAE stimulation
OAE measurement: reproducibility (%) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (otoacoustic emissions) which will take 2 minutes.
  Reproducibility during OAE stimulation
OAE measurement: respone level (dB SPL) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (otoacoustic emissions) which will take 2 minutes.
  "Amplitude" of the OAE response
OAE measurement: noise level (dB SPL) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (otoacoustic emissions) which will take 2 minutes.
  "Amplitude" of the noise level
OAE measurement: signal to noise ratio (dB) | This parameter will be assessed once during one of both testmoments (the motor/vestibular appointment), and is an outcome parameter of the hearing assessment (otoacoustic emissions) which will take 2 minutes.
  "Amplitude" of the noise level vs "amplitude" of the OAE response

CONTACTS AND LOCATIONS:
Overall Officials: Leen Maes, PhD, Principal Investigator — Ghent University and Ghent University Hospital
Locations (1):
- Ghent University, department rehabilitation sciences, Ghent, Belgium

REFERENCES:
- [Derived] Van Hecke R, Deconinck FJA, Wiersema JR, Clauws C, Danneels M, Dhooge I, Leyssens L, Van Waelvelde H, Maes L. Balanced Growth project: a protocol of a single-centre observational study on the involvement of the vestibular system in a child's motor and cognitive development. BMJ Open. 2021 Jun 11;11(6):e049165. doi: 10.1136/bmjopen-2021-049165. PMID 34117049